CLINICAL TRIAL: NCT04865211
Title: Does a ThoracoLumbar Interfacial Plane (TLIP) Block With Liposomal Bupivacaine Provide Extended Post-operative Analgesia Following Spinal Surgery
Brief Title: Does a ThoracoLumbar Interfacial Plane (TLIP) Block With Liposomal Bupivacaine Provide TLIP Block in Spinal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol #20-570
Record Dates: First submitted 2021-04-05; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative
Keywords: thoracolumbar; spine; pain; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Liposomal Bupivicaine (Experimental): Administration of a combination of lioposomal bupivicane 20ml/266mg mixed with 20mL of 0.375% bupivicaine
  Interventions: Drug: Liposomal bupivacaine
- Bupivicane (Active Comparator): Administration of 40 ml of 0.375% Bupivicaine with epinephrine 1:400,000
  Interventions: Drug: Bupivacaine Injection
- Placebo (Placebo Comparator): Saline injection with 40mL preservative-free saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liposomal bupivacaine — Use of liposomal bupivicaine as intraoperative local anesthesia
  Arms: Liposomal Bupivicaine
Drug: Bupivacaine Injection — Use of bupivicaine as intraoperative local anesthesia
  Arms: Bupivicane
Drug: Placebo — Use of saline as placebo for local anesthesia
  Arms: Placebo

SUMMARY:
The investigators are looking to recruit patients into a study demonstrating the effectiveness of a superficial nerve block involving the thoracolumbar interfascial plane (TLIP) in reducing postoperative pain in those undergoing spinal surgery

DETAILED DESCRIPTION:
Patients undergoing spine surgery with or without fusion experience a great deal of pain especially in the first 3 days after surgery. Spine surgeons are looking for ways to reduce the pain that you experience. Anesthesiologists have introduced a procedure, called a "TLIP block" to provide pain relief. The block involves injecting local anesthetic (numbing pain medication) in the lower back around the site of the surgery. This block has been used by other surgeons for other types of surgeries in the past and has been shown to work.

To determine how effective the block is, the investigators are conducting this investigational study where pain severity in patients who receive one of 2 kinds of local anesthetic or placebo are compared

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing multilevel lumbar spine surgery, age 18-75

Exclusion Criteria:

* Opioid use disorder, previous spine surgery, non english-speaking patients, patients with anticipated communication disorders, patients with coagulopathy, prisoners, children, pregnant women, single level hemilaminectomy with or without discectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-02-17 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in postoperative pain | 24-48 hours
  Using Visual Analog Scales on a scale of 0-10, where 0 is no pain and 10 is the worst pain
Total postoperative opioid requirements | 1-5 days
  Using daily MME

SECONDARY OUTCOMES:
Time to Ambulation | 1-5 days
  Daily physical therapy evaluations where ambulation is recorded and time from surgery is documented
Length of Hospital Stay | 1-5 days
  Number of postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Ueshima H, Hara E, Otake H. RETRACTED: Thoracolumbar interfascial plane block provides effective perioperative pain relief for patients undergoing lumbar spinal surgery; a prospective, randomized and double blinded trial. J Clin Anesth. 2019 Dec;58:12-17. doi: 10.1016/j.jclinane.2019.04.026. Epub 2019 Apr 25. PMID 31029989 (Retraction: PMID 35393187 J Clin Anesth. 2022 Aug;79:110690)
- [Background] Chen K, Wang L, Ning M, Dou L, Li W, Li Y. Evaluation of ultrasound-guided lateral thoracolumbar interfascial plane block for postoperative analgesia in lumbar spine fusion surgery: a prospective, randomized, and controlled clinical trial. PeerJ. 2019 Oct 28;7:e7967. doi: 10.7717/peerj.7967. eCollection 2019. PMID 31681518
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600